CLINICAL TRIAL: NCT00006485
Title: An Open-Labeled, Non-Randomized Phase I Study Of Flavopiridol Administered With Irinotecan (CPT-11) In Patients With Advanced Solid Tumors
Brief Title: Flavopiridol and Irinotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068316; MSKCC-00091; NCI-2272
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2003-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — alvocidib; Irinotecan

INTERVENTIONS:
Drug: alvocidib
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining flavopiridol with irinotecan in treating patients who have locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of flavopiridol when combined with irinotecan in patients with advanced solid tumors.
* Determine the clinical pharmacokinetics of this regimen, as well as the plasma levels of the active metabolite SN-38 and metabolic product SN-38 glucuronide in these patients.
* Determine, in a preliminary manner, the therapeutic activity of this regimen in these patients.
* Determine the role of p21 relative to treatment response and apoptosis in these patients treated with this regimen.

OUTLINE: This is a dose-escalation, open-label, non-randomized study of flavopiridol.

Patients receive irinotecan IV over 30 minutes followed 7 hours later by flavopiridol IV over 1 hour on days 1, 8, 15, and 22. Treatment continues every 6 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. During the first week of the second course, patients receive flavopiridol alone on day 1 and irinotecan alone on day 2.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients in the initial cohort experience dose limiting toxicity during the first course of treatment. An additional 10 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 44-50 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven locally advanced or metastatic solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Eligible for treatment at the maximum tolerated dose only if disease accessible for tissue biopsy by Tru-Cut, CT guidance, or endoscopy

  * Pleural effusions or abdominal ascites do not constitute adequate tissue for biopsy
* No known CNS metastasis or primary CNS tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Total neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT and SGPT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No cardiac arrhythmias, congestive heart failure, or myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing (during and for at least 2 months after study)
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after study
* No concurrent serious or uncontrolled infection
* HIV negative
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior irinotecan allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* No other concurrent investigational medication
* No concurrent vitamins (except a single multivitamin tablet), antioxidants, or herbal preparations or supplements
* No concurrent subcutaneous heparin or heparinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States